CLINICAL TRIAL: NCT07268547
Title: Wrist Reduction Intervention: Supracondylar Technique for Radial Nerve Block vs. Hematoma Block (WRIST Block Study)
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Sarasota Memorial Health Care System (Other)
Responsible Party: Principal Investigator, Aaron Grossberg, Principal Investigator, Sarasota Memorial Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-MEDI-58
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Wrist Fracture
Keywords: wrist fracture; fracture; nerve block
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to compare different types of local anesthesia-a supracondylar radial nerve block, a hematoma block, or a combination of the two-for lowering pain in people with a broken wrist (distal radius fracture). We want to find out which method provides better pain relief after the injury and during treatment in the emergency room. Each of these methods is a different standard procedure for pain control prior to wrist fracture reduction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Supracondylar radial nerve blocks (Experimental): Lidocaine injection given near the radial never under ultrasound guidance
  Interventions: Procedure: Supracondylar radial nerve block
- Hematoma blocks (Experimental): Injecting analgesia into the hematoma that forms surrounding the wrist fracture
  Interventions: Procedure: Hematoma block
- Combination of supracondylar radial nerve block and hematoma block (Experimental): Supracondylar radial nerve block given first followed by hematoma block
  Interventions: Procedure: Combination of blocks

INTERVENTIONS:
Procedure: Supracondylar radial nerve block — Supracondylar radial nerve blocks given at the radial nerve not as the same location of the fracture site, prior to fracture reduction.
  Arms: Supracondylar radial nerve blocks
Procedure: Hematoma block — Injection of analgesia into the hematoma that forms surrounding the wrist fracture.
  Arms: Hematoma blocks
Procedure: Combination of blocks — Supracondylar radial nerve block given first, followed by hematoma block, before fracture reduction.
  Arms: Combination of supracondylar radial nerve block and hematoma block

SUMMARY:
The purpose of this study is to compare different types of local anesthesia-a supracondylar radial nerve block, a hematoma block, or a combination of the two-for reducing pain in people with a broken wrist (distal radius fracture). This is being done to find out which method provides better pain relief after the injury and during treatment in the emergency room.

DETAILED DESCRIPTION:
This study is testing different ways to provide pain relief before reducing a broken wrist. Participants will receive one of three techniques: (1) a nerve block where a doctor injects lidocaine near the radial nerve under ultrasound guidance; (2) a hematoma block where a doctor injects lidocaine into the area where the bone broke; or (3) both the nerve block and the hematoma block. Patients will be asked how much pain they feel before the numbing, after the numbing, and after the wrist is reduced.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients admitted to the ECC with a distal radius fracture requiring closed reduction
* Patient must be willing and able to provide informed consent to the study

Exclusion Criteria:

* Under 18 years of age
* Pregnant
* Prisoner
* Allergy to lidocaine
* Patients unable to provide informed consent and/or perform study-related activities
* Patients undergoing procedural sedation
* Patients may be excluded at the discretion of the investigator based on their clinical judgment, if the participant no longer meets criteria, and/or if the health or safety of the patient may be impacted by taking part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain levels comparison | Pain will be measured at (1) baseline, (2) after administering the assigned pain block(s), and after the (3) fracture reduction.
  Comparing pain levels among patients who are undergoing a wrist fracture reduction. Measured on a scale of 0-10, 0= no pain to 10= worst pain.
  Pain will be measured at (1) baseline, (2) after administering the assigned pain block (s), and after the (3) fracture reduction.

SECONDARY OUTCOMES:
Amount of opioid medication needed to control pain. | Opioid medication prescribing will be assessed at baseline, time of admission to the emergency room, until the patient is discharged and they are no longer active in the study.
  The amount of opioid prescribed, if any, will be collected and recorded for comparison during patient's time in emergency room.
Number of patients requiring conscious sedation. | Patients will be monitored for need of conscious sedation from baseline, time of enrollment in the study, until discharge from the emergency room, when they are no longer active in the study.
  The need for conscious sedation among patients undergoing wrist fracture reduction in emergency care center will be recorded and monitored for comparison between groups.
Adverse Events Monitoring | From baseline, time the patient is admitted and enrolled into the study, until the patient is discharged and no longer active in the study.
  Adverse events associated with any of the blocks that are administered to patients undergoing a wrist fracture reduction in the emergency care center will be identified, monitored, and recorded for reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Grossberg, DO, Principal Investigator — Sarasota Memorial Health Care System
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tseng PT, Leu TH, Chen YW, Chen YP. Hematoma block or procedural sedation and analgesia, which is the most effective method of anesthesia in reduction of displaced distal radius fracture? J Orthop Surg Res. 2018 Mar 27;13(1):62. doi: 10.1186/s13018-018-0772-7. PMID 29580286
- [Background] Siebelt M, Hartholt KA, van Winden DFM, Boot F, Papathanasiou D, Verdouw BC, de Vries MR, Mathijssen NM, Kraan GA. Ultrasound-Guided Nerve Blocks as Analgesia for Nonoperative Management of Distal Radius Fractures-Two Consecutive Randomized Controlled Trials. J Orthop Trauma. 2019 Apr;33(4):e124-e130. doi: 10.1097/BOT.0000000000001388. PMID 30893220
- [Background] Oakley B, Busby C, Kulkarni S, Arnold SJ, Kulkarni SS, Ollivere BJ. Manipulation of distal radius fractures: a comparison of Bier's block vs haematoma block. Ann R Coll Surg Engl. 2023 May;105(5):434-440. doi: 10.1308/rcsann.2022.0116. Epub 2022 Oct 14. PMID 36239973
- [Background] Maia GAS, Cunha JC, Feijo CQ, Leal DM, Moreira JJ, Herrero CFPDS. Radial Nerve Supracondylar Block Versus Fracture Hematoma Block. Comparison of Their Efficacy in Cases of Fractures of the Distal Third of the Radius. Rev Bras Ortop (Sao Paulo). 2023 Aug 30;58(4):e557-e562. doi: 10.1055/s-0043-1768623. eCollection 2023 Aug. PMID 37663190
- [Background] Handoll HH, Madhok R, Dodds C. Anaesthesia for treating distal radial fracture in adults. Cochrane Database Syst Rev. 2002;2002(3):CD003320. doi: 10.1002/14651858.CD003320. PMID 12137688
- [Background] Haley CB, Beauchesne AR, Fox JC, Nelson AM. Block Time: A Multispecialty Systematic Review of Efficacy and Safety of Ultrasound-guided Upper Extremity Nerve Blocks. West J Emerg Med. 2023 Jun 30;24(4):774-785. doi: 10.5811/westjem.56058. PMID 37527380
- [Background] Gottlieb M, Cosby K. Ultrasound-guided hematoma block for distal radial and ulnar fractures. J Emerg Med. 2015 Mar;48(3):310-2. doi: 10.1016/j.jemermed.2014.09.063. Epub 2014 Dec 9. PMID 25497895
- [Background] Martinez-Arboleda JJ, Moreno M, Diaz-Solorzano JP, Mejia-Grueso A. Ultrasound-guided supracondylar radial nerve block for closed reduction of a distal radius fracture in the emergency department: Case report. Trauma Case Rep. 2024 Sep 25;54:101116. doi: 10.1016/j.tcr.2024.101116. eCollection 2024 Dec. PMID 39399762
- [Background] Che Daud AZ, Mohd Nayan NA, Ahmad A, Alrashdi M, Kadar M, Mohd Poot EF. Distal radius fracture rehabilitation: A bibliometric and scoping review. J Hand Ther. 2025 Jul 3:S0894-1130(25)00089-4. doi: 10.1016/j.jht.2025.05.016. Online ahead of print. PMID 40615307
- [Background] Abbasi S, Garjani N, Mahshidfar B, Farsi D, Mofidi M, Hafezimoghadam P, Rezai M, Javan A. Comparative Study of Radial and Median Nerve Blocks with Hematoma Block under Ultrasound Guide in Distal Radius Fracture Reduction: A Randomized Clinical Trial. Med J Islam Repub Iran. 2023 Oct 23;37:113. doi: 10.47176/mjiri.37.113. eCollection 2023. PMID 38145179